CLINICAL TRIAL: NCT01341522
Title: Clinical Evaluation of the Sorin Group's REPLY MR-conditional Pacing System
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IBMR01 - REPLY MRI STUDY
Record Dates: First submitted 2011-04-01; First posted 2011-04-25 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Dual-chamber Pacemaker Placement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Control
  Interventions: Procedure: control
- MRI (Experimental): experimental
  Interventions: Procedure: MRI exam

INTERVENTIONS:
Procedure: MRI exam — MRI exam
  Arms: MRI
Procedure: control — waiting room
  Arms: Control

SUMMARY:
Permanent cardiac pacemakers have represented a contraindication to Magnetic Resonance Imaging (MRI). Strong static, gradient and radiofrequency fields used for MRI are thought to be detrimental to pacemaker function and possibly cause harm to patients undergoing MRI examinations. A previous study has shown that MRI is indicated in 17% of all patients with pacemakers within 12 months of device placement , which demonstrates the need of practical, safe approach for performing MRI on pacemaker patients. A new Reply MR-conditional pacing system is developed by Sorin Group for safe use in the MRI environment. The new pacing system is composed by the Reply pacemaker and the Filtrea bradycardia pacing leads. This study intends to demonstrate the safety and the efficacy in the MRI environment of the Sorin Group Reply MR-conditional pacing system.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for dual-chamber pacemaker primo-implantation
* Patients who have indication for implantation of a dual-chamber pacemaker according to the American College of Cardiology and the American Heart Association
* Patients who are able and willing to undergo elective MRI scanning
* Patients who are scheduled for implant of a Reply DR pacemaker and Filtrea lead(s) only
* Patients who provided signed and dated informed consent

Exclusion Criteria:

* Non MR-compatible device or material implant
* Chronic atrial fibrillation (for atrial lead evaluation)
* Incessant ventricular tachyarrhythmia (for ventricular lead evaluation)
* Inability to understand the purpose of the study or refusal to co-operate
* Unavailability for scheduled follow-ups at the implanting centre
* Already included in another clinical study that could affect the results of this study
* Inability or refusal to provide informed consent
* Patient is minor (less than 18-year old)
* Patient is pregnant (women of childbearing potential should have a negative pregnancy test prior to enrolment);
* Patient has life expectancy of less than 1 year
* Patient is forfeiture of freedom or under guardianship
* Any patient to whom a contra-indication from device and lead labeling applies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
assess the pacing system-, MRI- and implant procedure-related complication-free rate | 1 month
assess atrial and ventricular lead-related complication-free rate | 3 months
compare the changes in atrial and ventricular pacing thresholds before and after MRI, between MRI and control groups | 3 months
compare the changes in atrial and ventricular sense amplitude after MRI between MRI and control groups | 3 months

SECONDARY OUTCOMES:
Summarize all implant procedure, pacing system- and MRI procedure-related adverse events | 12 months
Summarize atrial and ventricular electrical performances | 3 months
Summarize atrial and ventricular lead handling | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco LEYVA, Dr, Principal Investigator — Queen Elizabeth BIRMINGHAM UNITED KINGDOM